CLINICAL TRIAL: NCT00489593
Title: Phase I Dose-Finding Pilot Study of the Safety and Tolerability of Olanzapine in Patients With Advanced Cancer and Weight Loss
Brief Title: Olanzapine in Patients With Advanced Cancer and Weight Loss
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0620
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Advanced Cancer; Weight Loss
Keywords: Advanced Cancer; Weight Loss; Cachexia; Olanzapine; Zyprexa; Fluoxetine; Symbyax
MeSH Terms: conditions — Weight Loss; Cachexia | interventions — Olanzapine; Fluoxetine; olanzapine-fluoxetine combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Olanzapine (Experimental): Olanzapine 2.5 mg by mouth (PO) Daily x 28 days, increasing about every 3-14 days in increments of 2.5-5 mg until the designated dose for that cohort is reached.
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Olanzapine — 2.5 mg by mouth (PO) Daily x 28 days, increasing about every 3-14 days in increments of 2.5-5 mg until the designated dose for that cohort is reached.
  Other Names: Zyprexa; Fluoxetine; Symbyax

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of the drug Olanzapine that can be given to patients with advanced cancer who are experiencing weight loss. Researchers want to find out if Olanzapine can help decrease weight loss in patients who are experiencing it because of cancer. How this drug affects performance status, cancer-related symptoms, and nutritional status in patients with advanced cancer will also be studied.

DETAILED DESCRIPTION:
Olanzapine is approved for the treatment of schizophrenia and bipolar disorder. However, patients who have received this drug for these reasons have also experienced weight gain. Further studies in patients with cancer showed an improvement in appetite, a decrease in nausea, and a control of flushing (feeling of warmth) and sweating.

If you are found to be eligible to take part in this study and before you receive your first dose of Olanzapine, you will have routine blood tests (about 2 teaspoons). You will be asked a series of questions about your nutrition and how well you are able to perform daily activities. These questions should take about 20 minutes to answer. Your answers will help the study doctor decide if the study drug is helping you gain weight and if your weight gain is helping you feel better. You will also have an electrocardiogram (ECG - a test to measure the electrical activity of the heart). Women who are able to have children must have a negative blood pregnancy test (about 1 teaspoon).

After the tests above are completed, you will begin receiving Olanzapine. The study drug will be taken by mouth once daily at bedtime for 28 days in a row. Seven different doses of the drug are planned with 6 patients enrolled on each level. The level you are assigned to will depend on when you are enrolled on this study. All participants will begin taking the same strength of the study drug. This will gradually increase about every 3 - 14 days until you reach the highest strength of the study drug for the dose level to which you are assigned.

About every 2 weeks during this study for the first month and then about once a month thereafter, you will have a physical exam, including measurement of your vital signs (blood pressure, heart rate, temperature, and breathing rate), and your medical history will be discussed. You will also have routine blood tests (about 2 teaspoons) to check your general health.

You will continue to receive the highest strength of the study drug for the dose level to which you are assigned for about 4 months unless you have intolerable side effects or if your weight continues to decrease. The study doctor will decide if you should continue receiving Olanzapine after 4 months.

This is an investigational study. The FDA has approved Olanzapine for mental health diseases (schizophrenia, acute mania, and bipolar disorder). Its use in preventing weight loss is experimental. Up to 57 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with confirmed advanced cancer.
2. Patients with decreased daily caloric intake (<1500 Calories/day), or with a weight loss equivalent to 10% of body weight over six months
3. Patients should be able to have an oral intake and not be dependant on tube feeding, or have significant oropharyngeal obstruction, gastro-duodenal obstruction, or oral mucosal inflammation interfering with oral intake. Patients who have undergone gastro-jejunal bypass, esophagectomy, or total gastrectomy will be excluded.
4. ECOG performance status 2 or less.
5. Normal organ function: Creatinine less or equal to 2 times ULN; Bilirubin less or equal 2.5 times ULN
6. Ability to understand and the willingness to sign written informed consent.
7. Patients receiving concurrent chemotherapy or radiation therapy are eligible for enrollment.
8. Expected life expectancy of at least 3 months.

Exclusion Criteria:

1. Uncontrolled concurrent illness such as unstable angina, myocardial infarction in the preceding month, neutropenic fever, shock, symptomatic decompensate congestive heart failure, or congestive Heart Failure of NYHA III or IV, active internal bleeding.
2. Hypersensitivity to olanzapine, or history of dyskinesia or extrapyramidal syndrome on atypical neuroleptic.
3. Concurrent treatment with any atypical antipsychotic such as clozapine, risperidone, olanzapine, quetiapine, ziprasidone or aripiprazole
4. History of clozapine-induced agranulocytosis because patients will be at increased risk for neutropenia with Olanzapine.
5. Major surgery within four weeks of study start day.
6. Uncontrolled diabetes mellitus
7. Uncontrolled seizure disorder (any episode in the previous 4 weeks).
8. Pregnant and Nursing women.
9. Patients may not have started an appetite stimulant such as megace or therapeutic dose of steroids (superior or equal to an equivalent of 4 mg dexamethasone/day), or increased the dose of such medication (by more than 50%) in the previous week.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2006-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Toxicity evaluation after one 28-day cycle (& each dose level).

CONTACTS AND LOCATIONS:
Overall Officials: Aung Naing, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org